CLINICAL TRIAL: NCT07343193
Title: Deprescribing Antipsychotics: a Multiple Case Study
Acronym: DEPRESC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9822
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Psychotic Disorder
Keywords: Psychotic Disorder; Psychotic or Related Disorder; Antipsychotics
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The literature on antipsychotic deprescribing highlights the difficulty in establishing a clear consensus on the most optimal strategy due to the diversity of clinical situations encountered in daily practice: who should be deprescribed, when, at what rate, what strategy to employ in case of relapse, etc.

The fear of relapse leads psychiatrists (particularly in France) to tend to maintain long-term treatment, even if the arguments for this maintenance may be debatable due to an uncertain benefit-risk balance. Conversely, patients often request a reduction or discontinuation, notably because of the side effects of the treatments.

This argument serves to justify the value of presenting unique clinical situations like those in this study in a publication. The goal is for readers to gain a practical understanding of the successes and difficulties of deprescribing in real-life situations.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Patients with a psychotic or related disorder
* Patients on long-term antipsychotic treatment, clinically stable, who accept or request a deprescription between January 1, 2021, and October 30, 2025

Exclusion Criteria:

- Patients who have expressed their opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with a psychotic or related disorder
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Describe clinical situations where discontinuation of antipsychotics or a reduction of antipsychotics below the theoretically minimum recommended doses was possible. | Up to 12 months
  Stopping or reducing treatment:
  * Some patients may do well with less medication,
  * or even without medication, under carefully monitored conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie 1 - CHU de Strasbourg - France, Strasbourg, France